CLINICAL TRIAL: NCT05917327
Title: MEXWILS - Performance and Safety of MEX-CD1 Low-volume Continuous Veno-venous Haemodialysis Medical Device for Copper-extraction in Patients With Wilson's Disease
Brief Title: Performance and Safety of MEX-CD1 Low-volume Continuous Veno-venous Haemodialysis Medical Device for Copper-extraction in Patients With Wilson's Disease
Acronym: MEXWILS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Septex kit required has been discontinued by the external supplier
Sponsor: Mexbrain (Industry)
Collaborators: Integrated Scientific Services (ISS) AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJ2104-0003
Record Dates: First submitted 2023-04-06; First posted 2023-06-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Hepatolenticular Degeneration; Wilson
Keywords: Wilson's Disease; Low-volume continuous veno-venous hemodialysis; Copper
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective, multinational, multicentric, single-arm, open label, pivotal/registration clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MEX-CD1 Low volume CVVHD (Experimental): Patients enrolled in the treatment arm will receive MEX-CD1 treatment depending on the severity of their symptoms in addition to standard of care:
  * Patients with moderate liver injury not requiring extracorporeal blood epuration therapies as standard of care: 5 treatments with MEX-CD1 on consecutive days
  * Patients requiring extracorporeal blood epuration therapies as standard of care: 10 treatments with MEX-CD1 on consecutive days
  Interventions: Device: Low-volume continuous veno-venous haemodialysis

INTERVENTIONS:
Device: Low-volume continuous veno-venous haemodialysis — MEX-CD1 is a hyper-chelating colloidal solution that can be added to the dialysate to be used in low-volume continuous veno-venous hemodialysis. One treatment will last 4 hours. For non-hospitalized patients, the treatment is performed on an outpatient basis.

SUMMARY:
The goal of this clinical trial is to test the MEX-CD1 hemodialysis medical device in patients suffering from Wilson's Disease. The main questions it aims to answer are:

* Does the device work as expected by removing the excess of free copper from the blood?
* Is the device safe when used according to the instructions for use?

Depending on the severity of their symptoms, patients will receive either 5 or 10 treatments on consecutive days with the MEX-CD1 hemodialysis medical device.

DETAILED DESCRIPTION:
This study investigates the performance and safety of the MEX-CD1 hemodialysis device in patients suffering from Wilson's Disease. Wilson's Disease is a rare genetic disease (1'000 to 2'000 patients in France) linked to a problem in copper homeostasis. The direct consequence is a progressive accumulation of copper, first in the liver and then in the whole body with two major implications: (i) at the hepatic level and (ii) at the neurological level.

The disease is globally well known and managed in developed countries. It can present itself in several manners:

An acute decompensation of the disease is possible. This concerns mainly big children or young adults, presenting themselves with an acute hepatic deficiency that may need intensive care and a liver transplant.

In most cases, the clinical picture is one of chronic hepatic and/or neurological disease. Treatment must be adapted to the clinical situation. Two phases can be distinguished:

* A primary treatment phase, whose goal it is to eliminate the excess copper deposited in the body. This phase generally takes 1 to 2 years with chelating treatments;
* A maintenance phase, corresponding to the treatment which will allow the copper balance to be maintained and equilibrated.

This lifelong treatment is to be taken daily (with doses of chelators and/or zinc salts).

Finally, during the maintenance phase, periods of lesser observance or escape phases can be observed, those are responsible for severe aggravation of the liver (fulminant hepatitis) or of neurological symptoms that can lead to death.

The proposed medical device allows, by combining dialysis to a hyper-chelating colloidal dialysate (MEX-CD1) to specifically extract copper from the blood (and particularly the exchangeable copper). All patients enrolled in this study will, depending on the severity of their symptoms, receive 4-hour long treatments with MEX-CD1:

* Patients with moderate liver injury not requiring extracorporeal blood epuration therapies as standard of care: 5 treatments with MEX-CD1 on consecutive days
* Patients requiring extracorporeal blood epuration therapies as standard of care: 10 treatments with MEX-CD1 on consecutive days During the MEX-CD1 treatment, the patient's condition will be closely monitored. Additionally, enrolled patients will have a thorough assessment of their Wilson's Disease at the screening visit and at the last visit. Between the last day of treatment and the last visit, enrolled patients will have two rest days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 10 years and 80 years and weighing 30 kg and more
* Established diagnosis of Wilson disease (current Leipzig score ≥ 4). (For patients to whom Leipzig score can't be calculated at time of screening (while waiting for the genetic results), we assume a score of 4 (mutation detected on 2 chromosomes by default) if the two parents are Wilsonian.
* Adequate venous access to allow the setting up of recirculated low-volume continuous veno-venous hemodialysis (dialysis catheter ≥11.5 F, medium blood flow rate 100-200 mL/min) and the collection of blood samples.
* Both the patients already under Standard Of Care (SOC) or not under SOC.
* Patients must present at least one moderate hepatic or Neuropsychiatric symptom(s). (please refer 3.4 for the severity criteria)
* Patient, or parent or guardian in the case of minor, must have been informed about the nature of the clinical investigation, and must have agreed to participate in the clinical investigation, and signed the Informed Consent Form (ICF) prior to participation in any clinical investigation-related activities. Minors under the age of 14 must provide oral consent to participate in the clinical investigation.

Exclusion Criteria:

* Males and females weighing less than 30 kg
* Patients suffering from copper deficiency
* Patients who are unwilling or unable to comply with clinical investigation procedures
* Seafood allergy and prior allergy to one of the MEX-CD1 product components
* Allergy or contraindication to heparin or citrate
* Inadequate venous access
* Participation in another investigation with an investigational drug or another Medical Device (MD) within 30 days preceding, and during the present investigation
* Pregnant or breastfeeding women according to Article 66 of the Regulations (EU) 2017/745 on Medical Devices

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Performance of MEX-CD1 | 4 hours; from treatment start (0 hours) to treatment end (4 hours)
  The primary objective is to determine the performance of MEX-CD1 in terms of copper extraction in low-volume continuous veno-venous hemodialysis. This will be measured by the mean net amount of copper extracted per unit time relative to baseline, i.e., a proportion.

SECONDARY OUTCOMES:
Pulse measurement for safety purposes | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 2 weeks.
  Assessment of the safety of the MEX-CD1 medical device in low-volume continuous veno-venous hemodialysis. Safety end point measurements are evaluated throughout the study.
Temperature measurement for safety purposes | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 2 weeks.
  Assessment of the safety of the MEX-CD1 medical device in low-volume continuous veno-venous hemodialysis. Safety end point measurements are evaluated throughout the study.
Arterial blood pressure measurement every hour during treatment phase for safety purposes | Once at screening and last visit and every hour during treatment phase, assessed up to 2 weeks.
  Assessment of the safety of the MEX-CD1 medical device in low-volume continuous veno-venous hemodialysis. Safety end point measurements are evaluated throughout the study.
Weight measurement for Safety purposes | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 2 weeks.
  Assessment of the safety of the MEX-CD1 medical device in low-volume continuous veno-venous hemodialysis. Safety end point measurements are evaluated throughout the study.
  Weight measurement before and after each treatment.
AE recording | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 2 weeks.
  Assessment of the safety of the MEX-CD1 medical device in low-volume continuous veno-venous hemodialysis. Safety end point measurements are evaluated throughout the study.
Number of participants with abnormal laboratory test results | From the start of the first MEX-CD1 treatment until the last visit, assessed up to 2 weeks.
  Safety measurements via blood sample analysis before and after each 4-hour dialysis session
Responder rate | 4 hours; from treatment start (0 hours) to treatment end (4 hours)
  The responder rate is defined as the proportion of patients with >50% of the baseline net amount of exchangeable copper extracted throughout the study.
Copper kinetics | 4 hours; from treatment start (0 hours) to treatment end (4 hours)
  Kinetics of Copper measurement at time 0h, time 1h, time 2h, time 3h and time 4h
Changes in copper concentration between screening visit and last visit | Between the screening visit and the last visit, assessed up to 2 weeks.
  Assessment of the change in non-ceruloplasmin-bound copper (NCC) concentration between the baseline and the patient release
Hepatic function evolution | Between the screening visit and the last visit, assessed up to 2 weeks.
  Assessment of the stability or improvement of hepatic function between the enrolment and the last visit of the patient according to the history of the disease.
  Hepatic function is assessed through medical imaging, transient elastography (FibroScan or FibroTest), LiverMultiScan™, assessment of presence/absence of jaundice, assessment of presence/absence of haemolysis, ascites detection per sonography.
Neurologic and psychiatric status evolution | Between the screening visit and the last visit, assessed up to 2 weeks.
  Assessment of the stability or improvement of the neurological and psychiatric status between the enrolment and the last visit of the patient.
  Neurological and psychiatric status is evaluated with UWDRS scores, Clinical Global Impression-Improvement Scale (CGI-S versus CGI-I), MRI. (no units for all the scales)
Wilson's Disease evolution | Between the screening visit and the last visit, assessed up to 2 weeks.
  Assessment of the stability or improvement of the WD by Global Assessment Scale for WD between the enrolment and the last visit of the patient.

OTHER OUTCOMES:
non-ceruloplasmin-bound copper elimination and restoration during the treatment | 4 hours; from treatment start (0 hours) to treatment end (4 hours)
  Assessment of the non-ceruloplasmin-bound copper elimination and restoration along the dialysis session.
non-ceruloplasmin-bound copper restoration between treatment | End of treatment session (n) to beginning of next treatment session (n+1), assessed up to 2 weeks.
  Assessment of the non-ceruloplasmin-bound copper restoration between dialysis sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Edouardo COUCHONNAL-BEDOYA, Principal Investigator — Hôpital Femme Mère Enfant, Service Hépato-Gastroentérologie et Nutrition Pédiatrique
Locations (4):
- France (2):
  - Hôpital Femme Mère Enfant, Service des urgences et la réanimation pédiatriques, Bron, Auvergne-Rhône-Alpes
  - Hôpital Croix Rousse, Service d'hépatologie et gastroentérologie, Lyon, Auvergne-Rhône-Alpes
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Unitat de Trasplantament Hepàtic Pediàtric, Barcelona, Catalonia
  - Hospital Clinic Barcelona, Liver ICU, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No